CLINICAL TRIAL: NCT05947214
Title: Comparative Effects of Myofascial Decompression and Positional Release Therapies on Pain, Range of Motion and Functional Disability in Chronic Non-specific Neck Pain
Brief Title: Comparative Effects of Myofascial Decompression and Positional Release Therapies in Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0126
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: non-specific neck pain; myofascial decompression therapy; positional release therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Decompression Therapy (Experimental): 15 minute's moist heat will be given first. Patient was lied prone on couch with their upper torso unclothed, covered with massage oil than placed cup on skin and suction will created in cups by pump.
  Interventions: Other: Myofascial Decompression Therapy
- Positional Release technique (Experimental): Positional Release technique (PRT) is apply after application of moist heat pack for 15 minute. The subjects received PRT will be in supine lying with the therapist sitting on the affected side, tender points were located along with the upper fibers of trapezius muscle. The subject's head was laterally flexed towards the side of tender point, then therapist grasps the subject's forearm and abducts shoulder to approximately 900 and adds slight flexion or extension to fine-tune.
  Interventions: Other: positional Release Therapy

INTERVENTIONS:
Other: Myofascial Decompression Therapy — Group A will be given myofascial decompression therapy.15 minute's moist heat will be given first. Patient was lied prone on couch with their upper torso unclothed, covered with massage oil than placed cup on skin and suction will created by pump. Than drawn over skin along the spine from cervical to thoracic up to lateral border maintain the suction within skin throughout the procedure. The cup massage will conducted for approximately 10 minutes. Patients were informed that the treatment area may become patchy and there are chances of ecchymosis on the same area.
  Arms: Myofascial Decompression Therapy
Other: positional Release Therapy — Group B will be given Positional Release technique (PRT) after application of moist heat pack for 15 minute. The subjects received PRT will be in supine lying with the therapist sitting on the affected side, tender points were located along with the upper fibers of trapezius muscle. The subject's head was laterally flexed towards the side of tender point, then therapist grasps the subject's forearm and abducts shoulder to approximately 90 degree and adds slight flexion or extension to fine-tune. The ideal position of comfort achieved was held for a period of 90 sec and followed by passive return of body part to an anatomically neutral position continued for 5 minutes. Treatment duration was 3 sessions per week for 4 weeks.
  Arms: Positional Release technique

SUMMARY:
Nonspecific neck pain is defined as a neck pain not attributable to an identifiable, known specific pathology. The frequency of neck pain as found to be 84% which is exceptionally high and these are the majority of the individuals with neck pain that present to physiotherapy. In many cases, various factors contribute to the development of non-specific neck pain. These might include physical strain at work, such as working on something above you or sitting at a desk without moving enough. Emotional stress, like worries and anxiety about family or work, often plays an important role. It is thought that in some cases the cause may be an over-stretch (sprain) of a ligament or muscle. In other cases the cause may be a minor problem with a disc between two spinal bones (vertebrae), or a minor problem with a small facet joint between two vertebrae. Objective of this study will be to compare the effects of myofascial decompression and positional release therapies on pain, range of motion and functional disability in chronic nonspecific neck pain.

DETAILED DESCRIPTION:
Neck pain is one of the most common and painful musculoskeletal conditions. Point prevalence ranges from 6% to 22% and up to 38% of the elderly population, while lifetime prevalence ranges from 2% to 71%. For the majority of the neck disorders there is an absence of an identifiable underlying disease or abnormal anatomical structure. From this perspective .NS-NP is mainly 'diagnosed' on the basis of clinical grounds, provided there are no features to suggest a specific or more serious condition. The symptoms of nonspecific neck pain are similar to those of whiplash associated disorders (WAD) grade I and II but there is no traumatic event involved. Nonspecific neck pain (NP) is defined as pain in the posterior and lateral aspect of the neck between the superior nuchal line and the spinous process of the first thoracic vertebra with no signs or symptoms of major structural pathology and no or minor to major interference with activities of daily life as well as with the absence of neurological signs and specific pathologies. Chronic nonspecific neck pain is diagnosed as cervical pain without a known pathological basis as the underlying cause of the complaints. Some symptoms are limited cervical spine mobility and neck muscles weakness, which may be often related to other problems, such as, vertebral, neck or shoulder impaired function, and mental and physical stress at work. The natural course of non-specific neck pain remains unclear. While it is often self-limiting within a few weeks of onset, it can severely limit daily functioning, induce substantial medical consumption and result in prolonged sick leave and disability leading chronic nonspecific neck pain if pain duration is more than three months. As a consequence, it places a heavy burden on individuals, employers and health care services. Nonspecific neck pain is defined in the European guidelines for the management of chronic nonspecific neck pain that is not attributable to a recognizable, specific pathology (e.g., infection, tumor, osteoporosis, fracture, structural deformity, and inflammatory diseases, such as ankylosing spondylitis, radicular syndrome. Characteristic of chronic nonspecific neck pain are heavy pain, worsening with exertion and relieve with rest. In some cases the cause may be sprain or overstretch of a ligament or muscles. Nonspecific neck belongs to the group of musculoskeletal disorders, which include diverse conditions affecting muscles, bones, and/or joints of the limbs or the spine. As for most other musculoskeletal disorders, nonspecific neck is multifactorial. A variety of different types of exercise have been explored to treat chronic neck pain, including low-to-moderate intensity aerobic exercise, high intensity aerobic exercise, stretching exercise and muscular strength exercises and isometrics. However, the most effective form of exercise as a method of rehabilitation non-specific neck pain is unknown reflecting its complexity and more research is require. The rationale of the study is to compare the effects of myofascial decompression and positional release therapies on pain, range of motion and functional disability in chronic nonspecific neck pain. The main purpose of myofascial decompression therapy and positional release therapy is to release the cervical trigger points, improving end ranges and lengthening of muscle. MDT helps draw toxins out of the muscles and to the superficial veins to be removed by the body. This leads to decreased pain and tension in the tissues. The ultimate goal is to achieve pain free end ranges and flexibility of muscle in nonspecific neck pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Neck patients age 25 to 50 years.
2. Both male and female genders.
3. Mild to moderate back pain with NPRS pain score value of between more than 6/10.
4. Pain from at least past three months (12 weeks).
5. Trigger points within the muscle.

Exclusion Criteria:

1. Diagnosis of systemic metabolic and/or neurological disorders.
2. Patients with sensory impairments, such as diabetic sensory neuropathy. Neuropathic pain.
3. Any referred pain or neurological involvement in lower limbs is not included.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NPRS) | 6th week
  Numerical Rating Scale (NPRS) Numeric Rating Scale (NPRS) is most frequently used instruments to measure pain intensity in neck pain .The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
Neck Disability Index (NDI) | 6th week
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain. Points summed to a total score The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.,0 points or 0% means : no activity limitations .50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability. For patients' understanding, the URDU version is used. A clinically important change was calculated as 5 points, with a sensitivity of 0.78 and a specificity of 0.80

SECONDARY OUTCOMES:
ROM cervical spine (flexion) | 6th week
  The patient is seated with upper back supported with chair the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular or parallel to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor for measuring range of cervical flexion
ROM cervical spine (extension) | 6th week
  The patient is seated with upper back supported with chair the center of goniometer is placed over the external auditory meatus, proximal arm is Perpendicular or parallel to ground and distal arm With base of nares or parallel to longitudinal axis of tongue depressor and patient extend neck, for measuring the cervical extension ROM.
ROM cervical spine (side flexion) | 6th week
  The patient is seated with upper back supported with chair the center of goniometer is placed Over spinous process of C7,proximal arm over Spinous processes of thoracic vertebrae so that arm is perpendicular to ground and distal arm place over Dorsal midline of head. Reference occipital protuberance for side flexion
. ROM cervical spine (Rotation) | 6th week
  The patient is seated with upper back supported with a chair the center of the goniometer is placed Over center of cranial aspect of head, proximal arm is placed Parallel to imaginary line between the two acromial processes and distal arm With the tip of the nose. If using the tongue depressor, parallel to the longitudinal axis of tongue depressor for cervical rotation ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Hafeez, PhD*, Principal Investigator — Riphah International University Lahore Campus
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezzati K, Ravarian B, Saberi A, Salari A, Reyhanian Z, Khakpour M, Yousefzadeh Chabok S. Prevalence of Cervical Myofascial Pain Syndrome and its Correlation with the Severity of Pain and Disability in Patients with Chronic Non-specific Neck Pain. Arch Bone Jt Surg. 2021 Mar;9(2):230-234. doi: 10.22038/abjs.2020.48697.2415. PMID 34026942
- [Background] Rodriguez-Huguet M, Vinolo-Gil MJ, Gongora-Rodriguez J. Dry Needling in Physical Therapy Treatment of Chronic Neck Pain: Systematic Review. J Clin Med. 2022 Apr 23;11(9):2370. doi: 10.3390/jcm11092370. PMID 35566496
- [Background] Anwar S, Arsalan A, Zafar H, Ahmad A, Hanif A. Effects of breathing reeducation on cervical and pulmonary outcomes in patients with non specific chronic neck pain: A double blind randomized controlled trial. PLoS One. 2022 Aug 25;17(8):e0273471. doi: 10.1371/journal.pone.0273471. eCollection 2022. PMID 36006997
- [Background] Moustafa IM, Shousha TM, Walton LM, Raigangar V, Harrison DE. Reduction of Thoracic Hyper-Kyphosis Improves Short and Long Term Outcomes in Patients with Chronic Nonspecific Neck Pain: A Randomized Controlled Trial. J Clin Med. 2022 Oct 13;11(20):6028. doi: 10.3390/jcm11206028. PMID 36294349
- [Background] Peterson G, Peolsson A. Efficacy of Neck-Specific Exercise With Internet Support Versus Neck-Specific Exercise at a Physiotherapy Clinic in Chronic Whiplash-Associated Disorders: Multicenter Randomized Controlled Noninferiority Trial. J Med Internet Res. 2023 Jun 20;25:e43888. doi: 10.2196/43888. PMID 37338972
- [Background] Spellman J, Eldredge R, Nelson M, Ostrowski J, Concannon J. Is Myofascial Decompression Effective at Increasing Hamstring Flexibility in the Athletic Population? A Critically Appraised Topic. J Sport Rehabil. 2022 Aug 8;31(8):1100-1104. doi: 10.1123/jsr.2022-0013. Print 2022 Nov 1. PMID 35940580
- [Background] Parkinson SD, Zanotto GM, Maldonado MD, King MR, Haussler KK. The Effect of Capacitive-Resistive Electrical Therapy on Neck Pain and Dysfunction in Horses. J Equine Vet Sci. 2022 Oct;117:104091. doi: 10.1016/j.jevs.2022.104091. Epub 2022 Jul 29. PMID 35908601